CLINICAL TRIAL: NCT02374944
Title: A Randomized Clinical Trial Evaluating Fixation Insitu Versus Removal for Midfoot Lisfranc Injuries
Brief Title: Fixation Insitu Versus Removal for Midfoot Lisfranc Injuries
Acronym: FIRM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Calgary Orthopaedic Research and Education Fund (Other); Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Paul Duffy, Division Head, Orthopaedic Trauma, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB14-0625
Record Dates: First submitted 2015-02-10; First posted 2015-03-02 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Closed Fracture Dislocation, Tarsometatarsal Joint; Open Fracture Dislocation, Tarsometatarsal Joint
MeSH Terms: interventions — Hardware Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hardware Removal (Experimental): Removal of hardware at 6 months.
  Interventions: Procedure: Hardware removal
- Hardware Retention (No Intervention): Retention of hardware at 6 months

INTERVENTIONS:
Procedure: Hardware removal — Comparison of implant retention vs. scheduled implant removal in skeletally mature patients with previously operatively treated Lisfranc injuries requiring screw and/or plate fixation.
  Arms: Hardware Removal

SUMMARY:
This study is a multicenter prospective randomized control trial comparing hardware retention (HR) to removal of hardware (RH).

DETAILED DESCRIPTION:
Eligible patients will be randomized to one of two treatment arms: Hardware removal at 6 months or Hardware retention for a minimum of 2 years.

Consenting patients having previously undergone open reduction and internal fixation of Lisfranc injuries with an anatomic reconstruction within 6-8 weeks will be randomized to one of two treatment arms: removal hardware (RH) or hardware retention (HR).

Outcome will be assessed at 6 weeks, 12 weeks, 6 months, 1 year, and 2 years from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Subject has Lisfranc injury that was treated within 28 days of injury.
* Subject must be enrolled in study between 6 and 8 weeks from time of initial fixation operation.
* The patient must be medically fit for anesthesia
* Subject is willing and able to provide written informed consent for trial participation
* Subject is willing and able to comply with the study protocol including return for all follow-up evaluations
* Subject may have a bony, ligamentous, or combined lisfranc injury
* Demonstrated instability of the lisfranc complex on static, stress view or CT radiography.
* Associated injuries - other than the lisfranc complex - are permitted provided those injuries are not deemed to significantly influence the rehabilitation or recovery of the patient at the discretion of the enrolling surgeon
* Adequate reduction to within 1mm of lisfranc complex at time of fixation
* Hardware across the midfoot (tarsal-metatarsal joints 1-3)

Exclusion Criteria:

* Subject has a significant pre-existing foot injury
* Subject has a delay in initial treatment greater than 28 days from time of injury
* Subject has an active infection in the area of surgical approach requiring surgical debridement
* Subject has concomitant injury which, in the opinion of the attending surgeon, is likely to impair rehabilitation or prolong fracture healing time (another long bone fracture, ipsilateral limb injury)
* Subject has a history of rheumatoid arthritis, Diabetes, fibrous dysplasia, chronic renal failure, Paget's disease, or osteopetrosis or any other pre-existing pathologic condition affecting the Lisfranc complex
* Subject has a high risk of death from surgery (ASA physical status Class V)
* Subject is likely unable to maintain follow-up(no fixed address, plans to move out of town in the next year, states unable to comply with protocol, etc.)
* Subject has cognitive impairment or language difficulties that would impede the valid completion of questionnaires
* Subject is pregnant
* There has been loss of fixation or reduction prior to enrollment
* Previous corrective foot surgery
* Associated fracture of calcaneus, talus, or tibial plafond.
* Pathologic fracture
* Loss of fixation or reduction prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
AOFAS - American Orthopaedic Foot and Ankle Society Midfoot Score | 6 weeks
  Subjective and objective evaluation of the midfoot with breakdown by function (45 points), pain (40 points), and alignment (15 points) with a yield anywhere between 0 and 100 points where 100 points is a perfect score.
AOFAS - American Orthopaedic Foot and Ankle Society Midfoot Score | 12 weeks
  Subjective and objective evaluation of the midfoot with breakdown by function (45 points), pain (40 points), and alignment (15 points) with a yield anywhere between 0 and 100 points where 100 points is a perfect score.
AOFAS - American Orthopaedic Foot and Ankle Society Midfoot Score | 6 months
  Subjective and objective evaluation of the midfoot with breakdown by function (45 points), pain (40 points), and alignment (15 points) with a yield anywhere between 0 and 100 points where 100 points is a perfect score.
AOFAS - American Orthopaedic Foot and Ankle Society Midfoot Score | 1 year
  Subjective and objective evaluation of the midfoot with breakdown by function (45 points), pain (40 points), and alignment (15 points) with a yield anywhere between 0 and 100 points where 100 points is a perfect score.
AOFAS - American Orthopaedic Foot and Ankle Society Midfoot Score | 2 years
  Subjective and objective evaluation of the midfoot with breakdown by function (45 points), pain (40 points), and alignment (15 points) with a yield anywhere between 0 and 100 points where 100 points is a perfect score.
VAS-FA - Visual Analog Scale Foot and Ankle | 6 weeks
  Patient reported responses on 20 subjective questions (Pain - 4; functional deficits -13; other complaints - 3) equally weighted. Possible score out of 100.
VAS-FA - Visual Analog Scale Foot and Ankle | 12 weeks
  Patient reported responses on 20 subjective questions (Pain - 4; functional deficits -13; other complaints - 3) equally weighted. Possible score out of 100.
VAS-FA - Visual Analog Scale Foot and Ankle | 6 months
  Patient reported responses on 20 subjective questions (Pain - 4; functional deficits -13; other complaints - 3) equally weighted. Possible score out of 100.
VAS-FA - Visual Analog Scale Foot and Ankle | 1 year
  Patient reported responses on 20 subjective questions (Pain - 4; functional deficits -13; other complaints - 3) equally weighted. Possible score out of 100.
VAS-FA - Visual Analog Scale Foot and Ankle | 2 years
  Patient reported responses on 20 subjective questions (Pain - 4; functional deficits -13; other complaints - 3) equally weighted. Possible score out of 100.
SF-36 | 6 weeks
  Patient reported measure on physical and mental status on 36 items across eight health domains.
SF-36 | 12 weeks
  Patient reported measure on physical and mental status on 36 items across eight health domains.
SF-36 | 6 months
  Patient reported measure on physical and mental status on 36 items across eight health domains.
SF-36 | 1 year
  Patient reported measure on physical and mental status on 36 items across eight health domains.
SF-36 | 2 years
  Patient reported measure on physical and mental status on 36 items across eight health domains.
VAS - Visual Analogue Scale (Patient Satisfaction) | 6 weeks
  Single visual analogue scale to evaluate patient satisfaction on a scale of 0 to 100.
VAS - Visual Analogue Scale (Patient Satisfaction) | 12 weeks
  Single visual analogue scale to evaluate patient satisfaction on a scale of 0 to 100.
VAS - Visual Analogue Scale (Patient Satisfaction) | 6 months
  Single visual analogue scale to evaluate patient satisfaction on a scale of 0 to 100.
VAS - Visual Analogue Scale (Patient Satisfaction) | 1 year
  Single visual analogue scale to evaluate patient satisfaction on a scale of 0 to 100.
VAS - Visual Analogue Scale (Patient Satisfaction) | 2 years
  Single visual analogue scale to evaluate patient satisfaction on a scale of 0 to 100.

SECONDARY OUTCOMES:
Radiologic outcome | 2 years
  Radiographic measurement of the gap between 1st and 2nd metatarsals and maintenance of reduction on static and weight bearing xrays from index films at enrollment to 2 years.
Cost-effectiveness | 2 years
  Cost of treatment and complications plus incremental costs up to 2 year follow up will be collected and compared with Quality Adjusted Life Years (QALYs)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Duffy, MD, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - Foothills Medical Centre, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - South Health Campus, Calgary, Alberta